CLINICAL TRIAL: NCT00000176
Title: Alzheimer's Disease Prevention Trial. A Multi-center, Randomized, Double-blind Placebo Controlled Trial of Estrogens to Prevent Alzheimer's Disease and Loss of Memory in Women.
Brief Title: Alzheimer's Disease Prevention Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: IA0018; RO 1AG15922-01
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer Disease; Memory Disorders
Keywords: Alzheimer's disease; memory loss; Estrogen
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Estrogens; Progesterone

INTERVENTIONS:
Drug: Estrogen
Drug: Estrogen and Progesterone

SUMMARY:
This is a three-year study to determine if estrogens can prevent memory loss and Alzheimer's disease in women with a family history of Alzheimer's disease.

DETAILED DESCRIPTION:
PREventing Postmenopausal memory loss and Alzheimer's with Replacement Estrogens (PREPARE) is a double-blind-placebo controlled trial to determine whether estrogen (or estrogen and progesterone) can delay the onset of memory loss or Alzheimer's Disease in elderly women with a family history of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women 65 or older with a family history of memory problems not currently on estrogen.

Exclusion Criteria:

* Significant neurological impairment
* Current estrogen use
* History of breast cancer

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sano, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (22):
- United States (22):
  - University of Alabama, Birmingham, Alabama
  - University of California, Irvine, Irvine, California
  - New England Center for Headache, Stamford, Connecticut
  - Howard University, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Wein Center, Miami Beach, Florida
  - West Florida Regional Medical Center, Pensacola, Florida
  - North Broward Medical Center, Pompano Beach, Florida
  - Tallahassee Memorial Health Center, Tallahassee, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Columbia University, New York, New York
  - Cornell Medical Center, New York Presbyterian Medical Center, New York, New York
  - New York United Hospital Medical Center, Port Chester, New York
  - Burke Medical Research Institute, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Pharmaceutical Trials, Tulsa, Oklahoma
  - Butler Hospital, Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Background] Tang MX, Jacobs D, Stern Y, Marder K, Schofield P, Gurland B, Andrews H, Mayeux R. Effect of oestrogen during menopause on risk and age at onset of Alzheimer's disease. Lancet. 1996 Aug 17;348(9025):429-32. doi: 10.1016/S0140-6736(96)03356-9. PMID 8709781
- [Background] Kawas C, Resnick S, Morrison A, Brookmeyer R, Corrada M, Zonderman A, Bacal C, Lingle DD, Metter E. A prospective study of estrogen replacement therapy and the risk of developing Alzheimer's disease: the Baltimore Longitudinal Study of Aging. Neurology. 1997 Jun;48(6):1517-21. doi: 10.1212/wnl.48.6.1517. PMID 9191758
- [Background] Jacobs DM, Tang MX, Stern Y, Sano M, Marder K, Bell KL, Schofield P, Dooneief G, Gurland B, Mayeux R. Cognitive function in nondemented older women who took estrogen after menopause. Neurology. 1998 Feb;50(2):368-73. doi: 10.1212/wnl.50.2.368. PMID 9484355
- [Result] Aloysi A, Van Dyk K, Sano M. Women's cognitive and affective health and neuropsychiatry. Mt Sinai J Med. 2006 Nov;73(7):967-75. PMID 17195882